CLINICAL TRIAL: NCT00668018
Title: An Open-label, Multicenter Study to Assess Safety, Tolerability, Efficacy and Impact on Quality of Life of Vardenafil 10mg in Patients With Erectile Dysfunction Within a Time Window of up to 6 Hours After Intake of Study Drug
Brief Title: Assess Efficacy of Vardenafil 10mg in Erectile Dysfunction Within Intake of 6 Hours
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10678
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Male Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10mg orally on demand prior to intercourse

SUMMARY:
Assess efficacy of vardenafil within 6 hours after intake

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Males with erectile dysfunction
* Stable heterosexual relationship

Exclusion Criteria:

* Primary hypoactive sexual desire- History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Nitrate use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2003-01; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Successful attempt rate reported between drug ingestion and a maximum of 6 hours after drug intake | 12 weeks

SECONDARY OUTCOMES:
International Index of Erectile Function | 12 weeks
Global Assessment Question (GAQ) | 12 weeks
Other diary responses | 12 weeks
General Safety | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer